CLINICAL TRIAL: NCT03743844
Title: Compassion-focused Intervention for Women With Mood Disorders Seeking Treatment for Obesity
Brief Title: Psychosocial Intervention for Women With Mood Disorders Seeking Treatment for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Wharton Medical Clinic (Unknown); Women's College Hospital (Other)
Responsible Party: Principal Investigator, Dr. Eva Pila, Assistant Professor, University of Western Ontario, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0075-E
Record Dates: First submitted 2018-10-29; First posted 2018-11-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Mood Disorders
Keywords: weight management; compassion-focused treatment; internalized weight bias; depressive symptoms
MeSH Terms: conditions — Obesity; Mood Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion-focused psychoeducation group (Experimental): Receiving 2-hours of group-based in-person psychoeducational sessions weekly for 6-weeks.
  Interventions: Behavioral: Compassion-focused psychoeducation group
- Control group (No Intervention): Weight management treatment as usual

INTERVENTIONS:
Behavioral: Compassion-focused psychoeducation group — Attending six 2-hour weekly group-based psychoeducation sessions and participating in mindfulness, meditation, and acceptance-based experiential exercises
  Arms: Compassion-focused psychoeducation group

SUMMARY:
Women with mood disorders are vulnerable to the negative consequences associated with obesity, and face considerable challenges with adherence to behavioral weight management interventions. Strategies are needed to support the psychological well-being of this population, and improve adherence to weight-related treatment. The goal of this preliminary study is to determine the acceptability of a group-based compassion-focused psychoeducational intervention among women with mood disorders who are attending a behavioral weight management program.

DETAILED DESCRIPTION:
Pilot feasibility trial to examine the acceptability and efficacy of compassion-based intervention in reducing indices of psychopathology (i.e., internalized weight stigma, mood symptoms), and improving weight management outcomes (i.e., physical activity behaviour, dieting behaviour, weight loss) among women with mood disorders undergoing lifestyle weight management. In this proof of concept study, adult females with a diagnosis of major depressive disorder of bipolar disorder will be randomized into two arms: weight management treatment as usual + psychoeducation group; weight management as usual + control.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent form. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English.
* Female participants 18 - 65 years of age, inclusive, at the time of screening.
* Available and able to attend weekly group meeting on assigned dates.
* Diagnosis of major depressive disorder or bipolar disorder by a physician within the past 12 months, as indicated in WMC medical records and confirmed by MINI.
* Actively pursuing lifestyle weight management at WMC, with evidence of booked follow-up appointment.
* Weight status of at least 25kg/m2, as indicated by data from last appointment at WMC.
* Access to a computer and email account in order to complete online questionnaires

Exclusion Criteria:

* Enrolled in surgical management of obesity at WMC.
* Active substance abuse/dependence disorder, current suicidality, or active episode of psychosis.
* Presence of a hearing or visual impairment that will prevent completing the online surveys and from participating in a group discussion weekly meeting

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment from community-based clinic | 7-months (from baseline to 6-month follow-up)
  Proportion of eligible participants who agree to participate in the study
Adherence to the 6-week intervention | 6 weeks (from baseline to end of treatment)
  Proportion of sessions attended, and minutes spent weekly on home practice exercises

SECONDARY OUTCOMES:
Changes in internalized weight bias | 7 months (from baseline to 6-month follow-up)
  Weight Bias Internalization Scale (measures internalization of weight bias; mean score calculated, and ranges from 1 to 7)
Changes in depressive symptoms | 7 months (from baseline to 6-month follow-up)
  Beck Depression Inventory (measures depressive symptoms; total score calculated, and ranges from 0 to 63)
Changes in physical activity engagement | 7 months (from baseline to 6-month follow-up)
  International Physical Activity Questionnaire (measures physical activity frequency and intensity; continuous score of MET [Metabolic Equivalent Task] minutes per week)
Future adherence to weight management program | 7 months (from baseline to 6-month follow-up)
  Attending follow-up appointments

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No